CLINICAL TRIAL: NCT05383768
Title: Clinical Performance of Posterior Restorations of Bulk Fill Resin Composite Without Preheating Versus Repeated Preheating for One, Five and Ten Times: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Preheated and Repeated Preheated Versus Conventional Bulk Fill Resin Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Islam Ibrahim Mohammed, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20322
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Dental Leakage
MeSH Terms: conditions — Dental Leakage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Restoration with conventional no heated bulk-fill resin composite (Placebo Comparator): Restoration with conventional no heated bulk-fill resin composite, X-tra fill (VOCO, GERMANY)
  Interventions: Other: preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
- restoration with one-time preheated conventional bulk-fill resin composite (Active Comparator): restoration with one-time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
  Interventions: Other: preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
- restoration with five-time preheated conventional bulk-fill resin composite (Active Comparator): restoration with five-time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
  Interventions: Other: preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
- restoration with ten-time preheated conventional bulk-fill resin composite (Active Comparator): restoration with ten-time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C
  Interventions: Other: preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C

INTERVENTIONS:
Other: preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C — Intervention 1: restoration with one-time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C (Yang et al., 2020).
  Intervention 2: Restoration with five time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C (Yang et al., 2020).
  Intervention 3: Restoration with ten time preheated conventional bulk-fill resin composite, X-tra fill (VOCO, GERMANY) at 68◦C (Yang et al., 2020).

SUMMARY:
A Randomized clinical trial to evaluate the clinical Performance of Posterior Restorations of Bulk Fill Resin Composite without Preheating Versus Repeated Preheating for One, Five and Ten times .The null hypothesis of this study is that there is no significant difference in clinical performance of the restoration during restoring posterior teeth when using bulk-fill without preheating and after repeated preheating for one , five and ten times in restoration of posterior teeth.

DETAILED DESCRIPTION:
Dental resin composites are widely used for adhesive restorative procedures nowadays due to the significant improvement in their physical and mechanical properties. However, volumetric shrinkage is still an inherent drawback of the polymerization of the resin matrix .

Preheating improves adaptation, polymerization shrinkage and degree of conversion without affect mechanical properties of resin composite restorations.

In clinical situation, composite resin syringe is repeatedly used for restoration of several cavities and if preheating is applied, this syringe will undergo several heating cycles so repeated preheating effect on composite resin should be tested.

Follow up Period will be 1 year , Evaluation will be done at 3,6,9 and 12 months .

ELIGIBILITY:
Inclusion Criteria:

* a)Inclusion Criteria of participants

  1. Patient age between (18-60) years old.
  2. Patient is capable of informed consent. 3-Patients with a high level of oral hygiene.

     b)Inclusion Criteria of teeth:

  <!-- -->

  1. vital teeth
  2. Carious molar teeth.

Exclusion Criteria:

* a)Exclusion criteria of participants

  1. Participants with general systematic illness.
  2. Experience with allergic reactions against any component of used materials.
  3. Concomitant participation in another research study.
  4. Patients receiving Orthodontic treatment.
  5. Pregnant or lactating females.
  6. patient with heavy Bruxism habits.

     b)Exclusion criteria of the teeth

  <!-- -->

  1. The tooth to be filled is an abutment tooth for a removable prosthesis.
  2. The tooth to be filled is periodontally involved (grade 2 or grade 3 mobile).
  3. Endodontically treated tooth.
  4. tooth with previous restoration
  5. Exposed tooth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
(marginal integrity) using Modified US Public Health Service Criteria (USPHS) | one year
  Clinical Evaluation of restoration (marginal integrity) using Modified US Public Health Service Criteria (USPHS)

SECONDARY OUTCOMES:
(Marginal discoloration, secondary caries and Postoperative Sensitivity) using Modified US Public Health Service Criteria (USPHS) | one year
  Clinical Evaluation of restoration (Marginal discoloration, secondary caries and Postoperative Sensitivity) using Modified US Public Health Service Criteria (USPHS)

CONTACTS AND LOCATIONS:
Locations (1):
- Islam Ibrahim Mohammed, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05383768/Prot_000.pdf